CLINICAL TRIAL: NCT05596006
Title: Efficacy of ASIMOMMY® Compared to Domperidone and Placebo in Increasing Breastfeeding: Randomized Single-Blind Controlled Trial in Indonesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Andini Juwan Prabandari, MD, MD, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KE/FK/0191/EC/2022
Record Dates: First submitted 2022-10-23; First posted 2022-10-27 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Breastfeeding Mothers
Keywords: breastmilk; domperidone; neonates; ASIMOMMY®; Poly Herbal Formulation
MeSH Terms: interventions — Domperidone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ASIMOMMY® (Experimental): Experimental:
  2 capsules of ASIMOMMY, orally one times daily from days 1 to 7
  Interventions: Drug: ASIMOMMY®
- Domperidone (Active Comparator): Domperidone capsule, one capsule, orally three times daily from days 1 to 7
  Interventions: Drug: Domperidon
- Placebo (Placebo Comparator): Identical 2 capsules of placeb, orally one times daily from days 1 to 7
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASIMOMMY® — ASIMOMMY 500 mg
  Arms: ASIMOMMY®
Drug: Domperidon — Domperidone capsule 10 mg
  Arms: Domperidone
Drug: Placebo — Capsules of placebo 500mg.
  Arms: Placebo

SUMMARY:
The purpose of this study is assess the efficacy of ASIMOMMY® in increasing breast milk production in postpartum mothers.

DETAILED DESCRIPTION:
Several traditional herbs have been used and is well known since a long time ago by Indonesian people to increase the production of breastmilk, such as Katuk leaves (Sauropus androgynous Folium), Fenugreek (Trigonella foenum-graceum), and Moringa leaves (Moringa oleifera Folium). These plants have been scientifically proven through preclinical and even clinical research. However, not many have been further developed as phytopharmaceuticals that can be used in formal health services.

In previous research, ASI MOMMY® capsules have been successfully produced in accordance to the traditional method of making good herbal drugs, with each capsule containing extracts of Katuk leaf (300 mg), Fenugreek (150 mg), and Moringa leaf (50 mg). This formulation has gone through pharmacodynamic activity test, and acute and subactute toxicity test. Research has shown that ASI MOMMY® is works actively as a galactogogue and is not toxic, therefore it is safe to be given to humans (unpublished),

No research has been done to test the benefits of ASI MOMMY® in increasinng breastmilk production. Therefore, this research is a clinical trial that intends to see the benefits of ASI MOMMY® for increasing breastmilk production in postpartum women. This research is a part of the previous main research that is still ongoing to this day which aims to develop the formulation of ASI MOMMY® as a phytopharmaceutical

ELIGIBILITY:
Inclusion Criteria:

* Mothers 20-35 years old.
* Gestational age at delivery 37-40 weeks.
* Vaginal delivery.
* Normal body mass index (BMI 18.5-24.9 kg/m2).
* Not taking drugs or breast milk enhancement supplements.
* Healthy mother's condition with normal nipples (protruding).
* Healthy baby condition with good suction reflex.
* The baby consumes only breast milk.

Exclusion Criteria:

* Allergy to ASI MOMMY® and Domperidon.
* The mother is taking medications that affect the effects of domperidone (such as antacids, cimetidine, ranitidine, famotidine and nizatidine) or medications that interact with domperidone (such as haloperidol, lithium).
* The mother is in a state of illness requiring hospitalization.
* Mother has HIV AIDS, heart problems, mastitis, and had undergone breast surgery.
* Underweight, overweight and obese mothers.
* Giving birth to twins.
* The baby has a congenital defect that affects the suctioning process of breast milk
* Infants and mothers who did not participate in the treatment until completion (day 7 of the intervention).

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-12-31 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Increase in Neonates Weight | Day 0 to day 7
  The primary outcome is the difference in the neonates weight after 7 days of treatment with ASIMOMMY® compared to mothers receiving domperidone and placebo (mean day 7 neonates weight minus mean day 0 neonates weight).

SECONDARY OUTCOMES:
Proportion of non serious adverse event within 7 days | Day 0 to day 7
  Number of mothers or neonates who had non serious adverse event from day 0 to day 7 with ASIMOMMY® compare to mother receiving Domperidone and Placebo
Proportion of serious adverse event within 7 days | Day 0 to day 7
  Number of mothers or neonates who had serious adverse event from day 0 to day 7 with ASIMOMMY® compare to mother receiving Domperidone and Placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Health Center Jetis and Tegalrejo, Yogyakarta, DI Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT05596006/Prot_000.pdf
  • Informed Consent Form (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT05596006/ICF_001.pdf